CLINICAL TRIAL: NCT00005636
Title: A Single-Blind Randomized Phase III Trial of MTA Plus Cisplatin Versus Cisplatin in Patients With Malignant Pleural Mesothelioma
Brief Title: Cisplatin With or Without Pemetrexed Disodium in Treating Patients With Malignant Mesothelioma of the Pleura That Cannot be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 99-085; CDR0000067791 (Registry Identifier: PDQ (Physician Data Query)); CWRU-LILY-1599; LILLY-H3E-MC-JMCH(a); NCI-G00-1767
Record Dates: First submitted 2000-05-02; First posted 2004-05-26 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; Pemetrexed

INTERVENTIONS:
Drug: cisplatin
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if cisplatin is more effective with or without pemetrexed disodium for malignant mesothelioma of the pleura.

PURPOSE: Randomized phase III trial to compare the effectiveness of cisplatin with or without pemetrexed disodium in treating patients who have malignant mesothelioma of the pleura that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare survival in patients with malignant pleural mesothelioma when treated with cisplatin with or without LY231514. II. Compare duration of response, time to progression, and time to treatment failure in these patients with these treatment regimens. III. Compare tumor response rate and clinical benefit of these treatment regimens in these patients. IV. Compare Lung Cancer Symptom Scale scores, pulmonary function test scores, and lung density determinations with these treatment regimens in these patients. V. Compare toxicity of these treatment regimens in these patients. VI. Assess pharmacokinetics and vitamin metabolite status with these treatment regimens in these patients.

OUTLINE: This is a randomized, single blind, multicenter study. Patients are stratified according to performance status (Karnofsky 70-80% vs 90-100%), degree of measurability (bidimensional vs unidimensional only), histologic subtype (epithelial vs all others), WBC (8,300/mm3 and higher vs less than 8,300/mm3), pain intensity (low vs high), analgesic consumption (low vs high), dyspnea (low vs high), homocysteine (low vs high), gender, country, and treatment center. Patients are randomized to one of two treatment arms. Arm I: Patients receive LY231514 IV over 10 minutes followed by cisplatin IV over 2 hours on day 1. Arm II: Patients receive cisplatin as in arm I. Treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed at 4 weeks, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 280 patients (140 per treatment arm) will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant mesothelioma of the pleura not amenable to curative surgery Must be radiologically accessible Unidimensionally or bidimensionally measurable disease Pleural effusions or positive bone scan not considered measurable No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase, AST, and ALT no greater than 3.0 times ULN (no greater than 5 times ULN with liver involvement) Albumin at least 3.0 g/dL Renal: Creatinine clearance at least 45 mL/min Other: No serious systemic disorders that may preclude study No prior primary malignancy within the past 5 years except carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin No obvious malnourishment or greater than 10% weight loss within 6 weeks prior to study No active infection Not pregnant or nursing Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior immunomodulators allowed for pleurodesis No concurrent immunotherapy Chemotherapy: No prior systemic chemotherapy At least 1 week since prior bleomycin for pleurodesis Prior intracavitary cytotoxic drugs allowed for pleurodesis No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal anticancer therapy Radiotherapy: At least 4 weeks since prior radiotherapy to target lesion Lesion must be clearly progressive No concurrent radiotherapy Surgery: See Disease Characteristics No concurrent surgery for cancer Other: At least 4 weeks since any other prior investigational agent No concurrent aspirin or other nonsteroidal antiinflammatory drug from 2 days prior to 2 days after study (5 days prior for long acting agents such as piroxicam, naproxen, diflunisal, or nabumetone) No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ireland Cancer Center, Cleveland, Ohio